CLINICAL TRIAL: NCT05701189
Title: Phase 2, Randomized, Patient- and Rater-blinded Single-site Trial Evaluating Safety and Efficacy of Efgartigimod in Patients With Guillain-Barré Syndrome.
Brief Title: Evaluating Efgartigimod in Patients With Guillain-Barré Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chafic Karam (Other)
Collaborators: argenx (Industry)
Responsible Party: Sponsor-Investigator, Chafic Karam, Staff Physician and Associate Professor of Clinical Neurology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 852292
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — efgartigimod alfa; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod Alfa-Fcab (Experimental): 20mg/kg of Intravenous efgartigimod on days 1 and 5, with normal saline administered as placebo on days 2-4
  Interventions: Drug: Efgartigimod Alfa-Fcab
- Intravenous Immunoglobulin (IVIg) (Active Comparator): 0.4g/kg of IVIg daily for 5 days
  Interventions: Drug: Intravenous Immunoglobulin (IVIg)

INTERVENTIONS:
Drug: Efgartigimod Alfa-Fcab — Efgartigimod is an anti-neonatal Fc receptor (FcRn) immunoglobulin G1 Fc fragment. The FcRn plans a critical role in extending the half-life of IgGs by rescuing them from lysosomal degradation. Antibodies that bind and subsequently block the FcRn with high affinity result in IgGs being degraded more rapidly instead of salvaged. This approach has been shown to be beneficial in the antibody-mediated disorder myasthenia gravis.
  Other Names: Vyvgart
  Arms: Efgartigimod Alfa-Fcab
Drug: Intravenous Immunoglobulin (IVIg) — IVIg is the standard-of-care treatment for GBS. Brand of IVIG used may vary per institutional standards
  Other Names: Standard of Care IVIG
  Arms: Intravenous Immunoglobulin (IVIg)

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of Efgartigimod in patients with Guillain-Barre syndrome (GBS). The main questions it aims to answer are:

* Is Efgartigimod a safe treatment option for GBS patients?
* Does treatment with Efgartigimod improve patient outcomes?

In addition to standard-of-care procedures and assessments, participants will:

* Undergo seven blood draws during hospitalization and in four follow-up study visits to evaluate the concentration of neurofilament light chain, a protein that is elevated in patients with Guillain-Barré syndrome. The presence of neurofilament light chain is believed to be indicative of damage to the nervous system, with higher levels resulting from greater damage.
* Complete the Columbia Suicide Severity Rating Scale (C-SSRS) to monitor any suicidal ideation or behaviors during the course of the study.

DETAILED DESCRIPTION:
The following procedures/assessments are standard-of-care for Guillain-Barré syndrome. They will not be performed solely for research purposes in this study, but the study team will use select results from them to draw conclusions related to this research:

* The study doctor or study staff will ask you about your medical history and any changes to your medications
* You will have a physical examination
* Your vital signs, including blood pressure, pulse rate, breathing rate, body temperature, and weight will be measured
* You will have an electrocardiogram (ECG)
* Pulmonary function testing, including forced vital capacity (FVC), maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP) will be performed
* Blood samples will be drawn to evaluate disease progression and safety/efficacy of treatment
* You will undergo a lumbar puncture, commonly referred to as a spinal tap, to collect cerebrospinal fluid (CSF) for analysis
* Nerve conduction studies (NCS) will be performed
* Outcome assessments including the GBS Disability Scale (GBS-DS), MRC Sum Score, and Inflammatory Rasch-built Overall Disability Scale (I-RODS) will be performed

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 years or older
* Have a diagnosis of GBS according to the National Institute of Neurological Disorders and Stroke Diagnostic Criteria for Guillain-Barré Syndrome
* Onset of GBS-related weakness ≤14 days prior to infusion
* GBS-DS score of 3, 4, or 5

Exclusion Criteria:

* Pregnant and lactating women, and those intending to become pregnant during the trial or within 90 days after the last dosing. Women of childbearing potential should have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline prior to administration of IMP. Note: Women of childbearing potential should use a highly effective method of contraception (i.e., pregnancy rate of less than 1% per year) during the trial and for 90 days after the last administration of the IMP. They must be on a stable regimen, for at least 1 month, of combined estrogen and progestogen hormonal contraception with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or agree upon continuous abstinence from heterosexual sexual contact.
* Male patients who are sexually active and do not intend to use effective methods of contraception (as mentioned above) during the trial or within 90 days after the last dosing or male patients who plan to donate sperm during the trial or within 90 days after the last dosing. Note: Sterilized male patients who have had vasectomy with documented aspermia post-procedure, or male patients who have a partner of non-childbearing potential, can be included.
* GBS DS of 2 or less.
* Patients with any known severe bacterial, viral or fungal infection or any major episode of infection that required hospitalization or injectable antimicrobial therapy in the last 8 weeks prior to Screening.
* Patients with more than 14 days after onset of symptoms.
* Patients with known IgG deficiency.
* Patients with recurrent GBS.
* Use of investigational drug within 3 months or 5 half-lives of the drug (whichever is longer) prior to Screening.
* Patients who have a history of malignancy, including malignant thymoma, or myeloproliferative or lymphoproliferative disorders, unless deemed cured by adequate treatment with no evidence of recurrence for ≥ 3 years before Screening. Patients with completely excised non-melanoma skin cancer (such as basal cell carcinoma or squamous cell carcinoma) or cervical carcinoma in situ would be permitted at any time.
* Patients with clinical evidence of other significant serious disease or patients who underwent a recent major surgery, which could confound the results of the trial or put the patient at undue risk. Patients with renal/hepatic function impairment can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Guillain-Barre Syndrome Disability Scale (GBS-DS) | Week 4
  Scoring system that assesses the functional status of GBS subjects. Scores range from 0 to 6, with higher scores indicating a worse outcome.
Number and seriousness in adverse events in the studied population | Through study completion, an average of 3 years
  Safety monitoring

SECONDARY OUTCOMES:
Guillain-Barre Syndrome Disability Scale (GBS-DS) | 12 and 24 weeks
  Scoring system that assesses the functional status of GBS subjects. Scores range from 0 to 6, with higher scores indicating a worse outcome.
MRC Sum Score | 12 and 24 weeks
  Quantifies strength, with a higher score indicating more strength.
Inflammatory Rasch-Built Overall Disability Scale (I-RODS) | 4, 8, 12, and 24 weeks
  Functional outcome assessment. Scores range from 0 to 48, with higher scores indicating a better outcome.
Number of Days on Respirator | 4, 8, 12, and 24 weeks
  as noted in the title
Number of days in an intensive care unit | 4, 8, 12, and 24 weeks
  as noted in the title
Number of days to hospital discharge | 4, 8, 12, and 24 weeks
  as noted in the title
Mortality | 4, 8, 12, and 24 weeks
  Change in vital status
Percentage of patients with secondary deterioration due to treatment-related fluctuations (TRF) | 4, 8, 12, and 24 weeks
  as noted in the title
Adverse Events | 4, 8, 12, and 24 weeks
  occurrence of adverse events

OTHER OUTCOMES:
Study effect of Efgartigimod on IgG levels | change from baseline to 4 weeks and 24 weeks
  Blood sample to analyze change in IgG levels

CONTACTS AND LOCATIONS:
Overall Officials: Chafic Karam, MD, Principal Investigator — Staff Physician and Associate Professor of Clinical Neurology; Colin Quinn, MD, Study Director — Staff Physician and Associate Professor of Clinical Neurology
Locations (1):
- Hospital of University of Pennsylvania, Philadelphia, Pennsylvania, United States